CLINICAL TRIAL: NCT05986409
Title: The Role of Microbiota-gut-brain Axis as a Mediator in the Association Between Indoor Artificial Light at Night and the Relapse Risk of Schizophrenia: a Randomized, Crossover Trial
Brief Title: Indoor Artificial Light at Night and the Relapse Risk of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weizhuo Yi (Other)
Responsible Party: Sponsor-Investigator, Weizhuo Yi, Director, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20140101
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia Relapse; Light Pollution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opaque black tape covering part of the light source (Experimental): 10 wards were randomly selected as the intervention group (opaque black tape covering part of the light source).
  Interventions: Other: light cover
- no intervention (No Intervention): another 10 wards were selected as the control group (no intervention)

INTERVENTIONS:
Other: light cover — 10 wards were randomly selected as the intervention group (opaque black tape covering part of the light source), and another 10 wards were selected as the control group (no intervention).
  Arms: opaque black tape covering part of the light source

SUMMARY:
A randomized crossover trial of ALAN intervention was conducted in patients with chronic schizophrenia in Anhui Mental Health Center from August 15 to September 30, 2022. All participants met the diagnostic criteria for schizophrenia in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V). The enrolled patients were in the symptom-stable phase and were regularly prescribed antipsychotics (no change in medication regimen). The diets of all the participants were uniformly supplied during study. Patients with infectious diseases, eye diseases, or gastrointestinal diseases, or who used antibiotics at the time of recruitment, were excluded. The wards of the participants were all located in the same inpatient building. All included wards had the same size, layout, lighting and orientation of doors and windows. In normal conditions, each ward retains a small LED lamp (the same layout in all wards) at night as a source of lighting.

The study was divided into two stages. In the first stage, 10 wards were randomly selected as the intervention group (opaque black tape covering part of the light source), and another 10 wards were selected as the control group (no intervention). After a two-week washout interval, the second stage was carried out, with the two groups interchanging interventions. At the end of each intervention, participants completed a structured questionnaire scale to assess the relapse risk of schizophrenia, and then their fecal samples were collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Regularly taking antipsychotics

Exclusion Criteria:

* Infectious diseases
* Gastrointestinal diseases
* Using antibiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Relapse risk | up to 24 weeks
  Relapse risk was assessed by Chinese version of the Early Signs Scale (ESS). The ESS scale consists of 34 items (e.g., recently been bothered by 1 or 2 small things in life; To feel down and down; Other people don't understand me; Difficulty concentrating; It feels as if the thoughts are not my own... Etc.). Each entry is rated from 0 points (0 times/week), 1 score (1 time/week), 2 scores (more than 1 time/week) to 3 scores (at least 1 time/day), and all entries total 102 scores. The ESS scale has 4 dimensions, which are: Anxiety/agitation (ESS-A, 7 items); Depression/withdrawal (ESS - N, 10 items); Excitability/disinhibition (ESS-D, 6 items); Incipient psychosis (ESS-IP, 11 items).

SECONDARY OUTCOMES:
Cognitive function | up to 24 weeks
  The Montreal Cognitive Assessment (MoCA) is a widely used cognitive screening test designed to assess various cognitive functions, including memory, attention, language, and visuospatial abilities. It was created by Dr. Ziad Nasreddine in Montreal, Canada, in 1996, and it has since become a valuable tool for detecting mild cognitive impairment (MCI) and early signs of dementia, especially Alzheimer's disease.
  The MoCA consists of a series of tasks and questions that evaluate different cognitive domains. The total score on the MoCA is 30 points, with a higher score indicating better cognitive function. A score of 26 or above is considered normal for most individuals, although the normal range can vary based on factors such as age and education level.

CONTACTS AND LOCATIONS:
Overall Officials: Rubing Pan, Dr., Principal Investigator — Anhui Medical University
Locations (1):
- Weizhuo Yi, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No